CLINICAL TRIAL: NCT04519840
Title: A Cross Sectional Study to Determine the Association Between Diastasis Recti Abdominis and Sacroiliac Joint and Pelvic Floor Dysfunction Outcomes Among Postpartum Women Who Underwent C-section in UAE
Brief Title: Diastasis Recti Abdominis Association With Sacroiliac Joint and Pelvic Floor Dysfunction in Postpartum C-section Women
Status: Completed | Type: Observational
Sponsor: Dubai Health Authority (Other Government)
Responsible Party: Principal Investigator, Enas Mohammad Taher Abu Saleh, Physiotherapist, Dubai Health Authority
Other Study IDs: DubaiHA
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Diastasis Recti; Sacroiliac Joint Somatic Dysfunction; Pelvic Floor Disorders
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: nill — nill

SUMMARY:
Purpose: The purpose of the proposed study is to examine the ability of diastasis recti abdominis to predict outcomes of Sacroiliac joint dysfunction and pelvic floor dysfunction.

* Sample: The study will use a purposive sampling to select 120 subjects, ages 18-45, in the postpartum period between 12 weeks and 48 weeks. All subjects should have resided in the UAE minimum of 6 months prior to taking part in the study.

Data analysis:

* The age range of the subjects as well as the mean age with standard deviation will be determined.
* Data will be analyzed using Multivariate Linear Regression Analysis for the primary research question.
* For the Ssecondary research questions will include difference in DRA will be analyzed byas below:
* SIJ Dysfunction (logistic regression-Odds ratio)
* PFDI (Low, Moderate, High) (ANOVA/Kruskal Wallace Wallis Test)
* Pelvic Fascia excursion (Low, Moderate, High). (ANOVA/Kruskal Wallace Wallis Test)

DETAILED DESCRIPTION:
The data recorded for each subject will include: medical record number (MRN), type of delivery, measurement values and presence or absence of DRA as well as general health information collected in the health screening questionnaire. All identifiers will be kept separately , and password protected only accessed by Primary Investigator. Unless required by law or in the event of medical emergency, MRN of any subject will not be disclosed to anyone by the investigator. Under no circumstances will the personal identity of any subject be revealed in any form of a publication or presentation.

With the exception of the subject's medical record number as well as signed forms (consent and health questionnaire), all recorded study data will be identified using only a unique number for each subject. A paper master list will be kept that matches each medical record number to their identification number and kept in a separate locked and secured cabinet from the rest of the data. Other than that, the signed forms, all other data will be recorded initially on a paper sheet then transferred to an electronic spreadsheet. When not under direct supervision of the investigator, all paper records will be kept secure in locked filing cabinets, accessible only to the investigator. All data stored electronically will be maintained and backed up in an encrypted format with the password known only to the investigator. Subjects will be provided with a photocopy of the signed consent form.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participant should be 12-48 weeks postpartum between ages of 18-45 years
* Maximum two Cesarean section delivery with no vaginal deliveries.

Exclusion Criteria:

* ● Participant will be excluded (identified with the assistance of a health screening questionnaire):

  * History of traumatic injury to the lumbar-pelvic region, hip or lower extremities
  * Morbid Obesity: Participants with more than 35 kg/m2 body mass index will be excluded.
  * History of systemic disease affecting the musculoskeletal, neuromuscular and cardiopulmonary systems
  * Cardiovascular disease affecting lung function.
  * History of traumatic injury to the lumbar-pelvic region, hip or lower extremities.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — 12-48 weeks postpartum between ages of 18-45 years
Study Population: • The study will use a purposive sampling of 120 subjects, ages 18-45, in the postpartum period between 12 weeks and 48 weeks. All subjects will live in the United Arab Emirates minimum of 6 months prior to taking part in the study.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
presence of Diastasis Recti Abdominus | 48 weeks
  Primary outcome

SECONDARY OUTCOMES:
sacroiliac joint somatic dysfunction | 48 weeks
  Secondary outcome
Pelvic floor disorder | 48 weeks
  secondary outcome

CONTACTS AND LOCATIONS:
Overall Officials: Meeyoung Kim, PhD, Principal Investigator — University of Sharjah
Locations (1):
- Dubai Hospital, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
f prediction association is evident between diastasis recti abdominis and sacroiliac joint dysfuction medical record number and measurement scores will be used for further analysis for providing an experimental study. In which intervention will be applied for diastasis recti abdominis and observing the effect of that at sacroiliac joint dysfunction.
Supporting Information: ICF
Time Frame: one year
Access Criteria: only investigators

REFERENCES:
- [Background] Sperstad JB, Tennfjord MK, Hilde G, Ellstrom-Engh M, Bo K. Diastasis recti abdominis during pregnancy and 12 months after childbirth: prevalence, risk factors and report of lumbopelvic pain. Br J Sports Med. 2016 Sep;50(17):1092-6. doi: 10.1136/bjsports-2016-096065. Epub 2016 Jun 20. PMID 27324871
- [Background] Ostgaard HC, Roos-Hansson E, Zetherstrom G. Regression of back and posterior pelvic pain after pregnancy. Spine (Phila Pa 1976). 1996 Dec 1;21(23):2777-80. doi: 10.1097/00007632-199612010-00013. PMID 8979325
- [Background] Lee D, Hodges PW. Behavior of the Linea Alba During a Curl-up Task in Diastasis Rectus Abdominis: An Observational Study. J Orthop Sports Phys Ther. 2016 Jul;46(7):580-9. doi: 10.2519/jospt.2016.6536. PMID 27363572
- [Background] Vleeming A, Albert HB, Ostgaard HC, Sturesson B, Stuge B. European guidelines for the diagnosis and treatment of pelvic girdle pain. Eur Spine J. 2008 Jun;17(6):794-819. doi: 10.1007/s00586-008-0602-4. Epub 2008 Feb 8. PMID 18259783
- [Background] Broadhurst NA, Bond MJ. Pain provocation tests for the assessment of sacroiliac joint dysfunction. J Spinal Disord. 1998 Aug;11(4):341-5. PMID 9726305
- [Background] Laslett M, Aprill CN, McDonald B, Young SB. Diagnosis of sacroiliac joint pain: validity of individual provocation tests and composites of tests. Man Ther. 2005 Aug;10(3):207-18. doi: 10.1016/j.math.2005.01.003. PMID 16038856
- [Background] Vleeming A, de Vries HJ, Mens JM, van Wingerden JP. Possible role of the long dorsal sacroiliac ligament in women with peripartum pelvic pain. Acta Obstet Gynecol Scand. 2002 May;81(5):430-6. doi: 10.1034/j.1600-0412.2002.810510.x. PMID 12027817
- [Background] Freburger JK, Riddle DL. Using published evidence to guide the examination of the sacroiliac joint region. Phys Ther. 2001 May;81(5):1135-43. No abstract available. PMID 11319939
- [Background] O'Sullivan PB, Beales DJ, Beetham JA, Cripps J, Graf F, Lin IB, Tucker B, Avery A. Altered motor control strategies in subjects with sacroiliac joint pain during the active straight-leg-raise test. Spine (Phila Pa 1976). 2002 Jan 1;27(1):E1-8. doi: 10.1097/00007632-200201010-00015. PMID 11805650
- [Background] Bruno PA, Millar DP, Goertzen DA. Inter-rater agreement, sensitivity, and specificity of the prone hip extension test and active straight leg raise test. Chiropr Man Therap. 2014 Jun 16;22:23. doi: 10.1186/2045-709X-22-23. eCollection 2014. PMID 24982755
- [Background] Mota P, Pascoal AG, Sancho F, Bo K. Test-retest and intrarater reliability of 2-dimensional ultrasound measurements of distance between rectus abdominis in women. J Orthop Sports Phys Ther. 2012 Nov;42(11):940-6. doi: 10.2519/jospt.2012.4115. Epub 2012 Jul 18. PMID 22810966
- [Background] Chiarello CM, McAuley JA. Concurrent validity of calipers and ultrasound imaging to measure interrecti distance. J Orthop Sports Phys Ther. 2013;43(7):495-503. doi: 10.2519/jospt.2013.4449. Epub 2013 Apr 30. PMID 23633625
- [Background] Butowicz CM, Ebaugh DD, Noehren B, Silfies SP. VALIDATION OF TWO CLINICAL MEASURES OF CORE STABILITY. Int J Sports Phys Ther. 2016 Feb;11(1):15-23. PMID 26900496
- [Background] Barton A, Serrao C, Thompson J, Briffa K. Transabdominal ultrasound to assess pelvic floor muscle performance during abdominal curl in exercising women. Int Urogynecol J. 2015 Dec;26(12):1789-95. doi: 10.1007/s00192-015-2791-9. Epub 2015 Jul 28. PMID 26215905
- [Background] Fonseca H, Silva AM, Matos MG, Esteves I, Costa P, Guerra A, Gomes-Pedro J. Validity of BMI based on self-reported weight and height in adolescents. Acta Paediatr. 2010 Jan;99(1):83-8. doi: 10.1111/j.1651-2227.2009.01518.x. PMID 19878130
- [Background] Al-Shehri AH, Taha AZ, Bahnassy AA, Salah M. Health-related quality of life in type 2 diabetic patients. Ann Saudi Med. 2008 Sep-Oct;28(5):352-60. doi: 10.5144/0256-4947.2008.352. PMID 18779640
- [Result] Mota P, Pascoal AG, Carita AI, Bo K. Normal width of the inter-recti distance in pregnant and postpartum primiparous women. Musculoskelet Sci Pract. 2018 Jun;35:34-37. doi: 10.1016/j.msksp.2018.02.004. Epub 2018 Feb 20. PMID 29494833
- [Result] Bo K, Hilde G, Tennfjord MK, Sperstad JB, Engh ME. Pelvic floor muscle function, pelvic floor dysfunction and diastasis recti abdominis: Prospective cohort study. Neurourol Urodyn. 2017 Mar;36(3):716-721. doi: 10.1002/nau.23005. Epub 2016 Mar 31. PMID 27037746
- [Result] Gillard S, Ryan CG, Stokes M, Warner M, Dixon J. Effects of posture and anatomical location on inter-recti distance measured using ultrasound imaging in parous women. Musculoskelet Sci Pract. 2018 Apr;34:1-7. doi: 10.1016/j.msksp.2017.11.010. Epub 2017 Nov 22. PMID 29195217
- [Result] Mota P., Pascoal A.G., Vaz C., João F., Veloso A., Bø K. (2018) Diastasis Recti During Pregnancy and Postpartum. In: Brandão S., Da Roza T., Ramos I., Mascarenhas T. (eds) Women's Health and Biomechanics. Lecture Notes in Computational Vision and Biomechanics, vol 29. Springer, Cham. https://doi.org/10.1007/978-3-319-71574-2_10